CLINICAL TRIAL: NCT00483106
Title: Clinical and Pharmacogenetic Study of Attention Deficit With Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Ridha Joober, Md, PhD., McGill University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 99-22
Record Dates: First submitted 2007-06-04; First posted 2007-06-06 (Estimated); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; Genetics; Pharmacogenetics
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ritalin (Active Comparator)
  Interventions: Drug: Ritalin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ritalin — 0.25 mg/kg bid, orally for 7 consecutive days
  Arms: Ritalin
Drug: Placebo — taken orally twice a day for 7 consecutive days
  Arms: Placebo

SUMMARY:
Attention deficit with hyperactivity disorder (ADHD) is a very common behavioral problem during childhood. It is estimated that up to 80% of this disorder could be related to genetic factors. The most common treatment for ADHD is psychostimulants. In this study, the researchers investigate the effect of genetic variants in increasing the risk for behaviours pertinent to ADHD or in modulating the response of these behaviours to methylphenidate. Response to methylphenidate is evaluated through a double blind placebo controlled one week study.

DETAILED DESCRIPTION:
Attention Deficit Hyperactivity disorder (ADHD) is a syndrome that is characterized by inattention, motor hyperactivity and impulsivity. It affects 8 to 12% of the population. The presentation of children with ADHD can be varied, from simple inattention to severe motor hyperactivity and impulsivity. It has a negative impact on the child's life, including poor school achievement and difficulty with peer and family relationships.

Although the etiology of ADHD is not well understood, genetic factors are known to play a significant role in the pathogenesis of ADHD, as indicated by family, twin and adoption studies. In addition, environmental factors such as smoking during pregnancy and obstetrical complications have been found to contribute significantly in increasing the risk for and severity of ADHD. It is therefore likely that genetic predisposing factors interact with environmental factors to produce the behavioral disturbances observed in ADHD. The first goal of this study is therefore to investigate possible genetic and environmental risk factors, and examine how they might interact to confer increased risk for ADHD.

A majority of children (70%) with ADHD show a significant improvement with of their behavioral disorder when treated with stimulant drugs such as methylphenidate (MPH). However, the extent to which each child benefits from MPH is variable and some of the children do not improve at all in spite of adequate trials with stimulant drugs. The second purpose of this project is to study the correlates/predictors of responsiveness to MPH in school-aged children and to identify genetic factors that may modulate the behavioral response to this drug.

In order to achieve our research goals, children with ADHD are invited to participate to a two-week double-blind placebo controlled medication trial with MPH (Ritalin, 0.5mg/kg/day). During these two weeks, neuropsychological and behavioral assessments of the child are performed at the clinic to evaluate the cognitive performance of the child while on medication and placebo. Parents are invited to answer questionnaires about the behavior of their child and about family history of mental disorders, as well as prenatal and perinatal risk factors. Finally, the participating child, both parents, and siblings are invited to provide a blood or saliva sample for genetic analysis.

ELIGIBILITY:
Inclusion Criteria:

* ADHD

Exclusion Criteria:

* Psychosis
* Tourette syndrome
* Intelligence quotient (IQ) < 70
* Pervasive developmental disorder (PDD)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 885 (Actual)
Dates: Start 1999-11 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Conners' Global Index - Parent Version (CGI-P) | Once weekly during the medication trial
  10-item standardized scale evaluating ADHD symptoms; filled by parents.
Conner's Global Index - Teacher Version (CGI-T) | Once weekly during the medication trial
  10-item standardized scale evaluating ADHD symptoms; filled by teachers.

CONTACTS AND LOCATIONS:
Overall Officials: Ridha Joober, MD, PhD, Principal Investigator — Douglas Mental Health University Institute; Natalie Grizenko, MD, FRCPC, Principal Investigator — Douglas Mental Health University Institute
Locations (1):
- Douglas Mental Health University Institute, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Fageera W, Chaumette B, Fortier ME, Grizenko N, Labbe A, Sengupta SM, Joober R. Association between COMT methylation and response to treatment in children with ADHD. J Psychiatr Res. 2021 Mar;135:86-93. doi: 10.1016/j.jpsychires.2021.01.008. Epub 2021 Jan 7. PMID 33453563
- [Derived] Naumova D, Grizenko N, Sengupta SM, Joober R. DRD4 exon 3 genotype and ADHD: Randomised pharmacodynamic investigation of treatment response to methylphenidate. World J Biol Psychiatry. 2019 Jul;20(6):486-495. doi: 10.1080/15622975.2017.1410221. Epub 2017 Dec 15. PMID 29182037
- [Derived] Fageera W, Traicu A, Sengupta SM, Fortier ME, Choudhry Z, Labbe A, Grizenko N, Joober R. Placebo response and its determinants in children with ADHD across multiple observers and settings: A randomized clinical trial. Int J Methods Psychiatr Res. 2018 Mar;27(1):e1572. doi: 10.1002/mpr.1572. Epub 2017 Jun 30. PMID 28664541
- [Derived] Grizenko N, Cai E, Jolicoeur C, Ter-Stepanian M, Joober R. Effects of methylphenidate on acute math performance in children with attention-deficit hyperactivity disorder. Can J Psychiatry. 2013 Nov;58(11):632-9. doi: 10.1177/070674371305801109. PMID 24246434
- [Derived] Thakur GA, Sengupta SM, Grizenko N, Choudhry Z, Joober R. Comprehensive phenotype/genotype analyses of the norepinephrine transporter gene (SLC6A2) in ADHD: relation to maternal smoking during pregnancy. PLoS One. 2012;7(11):e49616. doi: 10.1371/journal.pone.0049616. Epub 2012 Nov 20. PMID 23185385
- [Derived] Thakur GA, Sengupta SM, Grizenko N, Choudhry Z, Joober R. Family-based association study of ADHD and genes increasing the risk for smoking behaviours. Arch Dis Child. 2012 Dec;97(12):1027-33. doi: 10.1136/archdischild-2012-301882. Epub 2012 Oct 29. PMID 23109089
- [Derived] Thakur GA, Grizenko N, Sengupta SM, Schmitz N, Joober R. The 5-HTTLPR polymorphism of the serotonin transporter gene and short term behavioral response to methylphenidate in children with ADHD. BMC Psychiatry. 2010 Jun 22;10:50. doi: 10.1186/1471-244X-10-50. PMID 20569447
- [Derived] Ter-Stepanian M, Grizenko N, Zappitelli M, Joober R. Clinical response to methylphenidate in children diagnosed with attention-deficit hyperactivity disorder and comorbid psychiatric disorders. Can J Psychiatry. 2010 May;55(5):305-12. doi: 10.1177/070674371005500506. PMID 20482957